CLINICAL TRIAL: NCT03398499
Title: Physiotherapeutic Rehabilitation to Eliminate Temporomandibular Joint Pain in Patients After Orthognathic Surgeries
Brief Title: Physiotherapeutic Rehabilitation in Patients After Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: Ministry of Health, Poland (Other Government)
Responsible Party: Principal Investigator, Edward Kijak, Principal Investigator, Pomeranian Medical University Szczecin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB-0012/149/15
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2018-01

CONDITIONS: TMJ Pain
Keywords: pain; orthognathic surgery; temporomandibular disorders (TMD); Electromagnetic Therapy; Light therapy
MeSH Terms: conditions — Pain; Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: Rehabilitation of patients after orthognathic procedures was performed, in which orthognathic surgery was performed - Bilateral Sagittal Split Osteotomy (BSSO). In the study it was used treatments a combination physicotherapies that combines two therapeutic physical factors - the electromagnetic field and the electromagnetic wave of red and infrared light in the form of led light therapy generated by the Viofor JPS device (Med&Life, Poland). Treatments with a slow-changing electromagnetic field were carried out using ring and elliptic applicators. Treatments with magnetoledotherapy using elliptical magnetic applicators combined with light. For physiotherapeutic purposes, led lighttherapy was used, which is a combined use of Extremely Low Frequency Magnetic Field (ELF-MF) and light coming from high energy LEDs (Light Emitting Diode) in the range of red (R) and infrared (IR). Therapies were used once a day, doing three described applications for a period of 10 days.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetoledotherapy (Experimental): Active ELF EMF Participants will receive active transcranial low frequency elec-tromagnetic field and magnetic induction (ELF EMF) and high energy LED light were used stimulation,Using the Viofor JPS device (Med & Live)
  Interventions: Device: VIOFOR (Med & Life)

INTERVENTIONS:
Device: VIOFOR (Med & Life) — Device: VIOFOR (Med & Life) Magnetic-light applicators, generating a slow-changing electromagnetic field and light ener-gy (830 nm and 640 nm), emitted from LEDs during a physiotherapeutic treatment application parameters: frequency of basic field pulses: 180-195 Hz frequency of packet the field pulses: 12.5 Hz-29 Hz magnetic induction: 15 μT wavelength of light: 830 nm and 640 nm Duration: 10 min number of treatments: 10
  Other Names: Combination physicotherapies; Magnetoledotherapy

SUMMARY:
Orthognathic surgery procedures are often used to correct for skeletal II and III skeletal deformation, dental-facial-maxillary deformation, mandibular laterognathy and maxillofacial asymmetry. The factors that motivate patients to undergo this procedure are: improvement of chewing, speech and swallowing as well as aesthetic and psychosocial factors. Correction of occlusal-facial defects requires team orthodontic, surgical and rehabilitation treatment. As with any surgical procedure, various preoperative, intraoperative and postoperative com-plications may occur. Late complications that may occur in variously long periods of time from surgery include among others dysfunction of the temporomandibular joint, idiopathic atrophy of the condyloid muscles and associated pain. After orthognathic operations, pain occurs almost always, although the degree of its severity is a subjective sensation of each patient. Regardless of intensity, the fight against pain is one of the basic activities in post-operative care of the patient. The aim of the study was to evaluate the effectiveness of the physiotherapeutic method, which uses a slow-changing electromagnetic field and light ener-gy emitted from high-energy LEDs - light emitting diode, Magnetholedoterpy, in reducing pain in patients after orthognathic surgery Using the Viofor JPS device (Med & Live)

DETAILED DESCRIPTION:
BACKGROUND:

Patients with dental-facial deformity require orthognathic surgery to improve face profile and asymmetry, and to correct malocclusion. Positional changes in the mandible, jaw or both jaws during can affect the temporomandibular joint (TMJ), chewing muscles, surrounding soft tis-sue and symptoms of joint dysfunction (TMD). Pain is a natural response of the body to injury and at the same time one of the symptoms defining the inflammatory reaction. Orthognathic surgery procedures are often used to correct skeletal deformation II and III of the skeletal class, dental-facial-maxillary deformation, mandibular laterognathion and maximal-facial asymmetry. After-care care of the patient aims to minimize the risk of complications and therapy of existing ones. Regardless of intensity, the fight against pain is one of the basic activities in post-operative care of the patient. Some studies have shown that patients undergo-ing physiotherapeutic care immediately recover from the surgery much more quickly. The use of physical treatments allows to obtain a significant faster improvement in the pain and associated swelling after surgery.

PROBLEM:

The motivating factors for patients undergoing orthognathic surgery are: improvement of chewing, speech and swallowing as well as aesthetic and psychosocial factors. Correction of occlusal defects requires a group orthodontic, surgical and rehabilitation treatment. Surgical techniques that have evolved over the last decades now allow for almost any displacement within the bony structures of the jaw and mandible. The pain after orthogonal surgery occurs almost always, although the degree of its severity is the subjective sensation of each patient. Patients above all experience pain from mild to severe. His post-operative treatment is very important to reduce the stress caused the occurrence itself pain. Postoperative pain is often controlled by the use of opioids, which are often used in the United States. Cold compresses are also used in the stimulus treatment to reduce pain related associated with the occurrence of edema. Regardless of intensity, the fight against pain is one of the basic activities in post-operative care of the patient. Pharmacotherapy often necessary also causes a number of adverse effects harmful to the whole organism. In order to restore the physical and psychological comfort of patients after orthognathic procedures, physiotherapeutic methods as well as physiotherapeutic devices can be used.

AIM:

The aim of the study was to assess the effectiveness of the combined physiotherapeutic method, which uses a slow-changing electromagnetic(ELF EMF) field and light energy, emitted from high-energy LEDs, in reducing pain in patients after orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19-24 years, both male and female
* Provide informed consent to participate in the study;
* Having a diagnosis of TMJ pain (TMD) according to RDC/TMD
* Visual analogic scale (VAS) score from 4 to 10 for 14 days
* Not pregnant;
* Not have contraindications to Extremely Low Frequency- Electro Magnetic Field(ELF EMF), such as implanted brain devices;
* Not have history of alcohol or drugs abuse within the past 6 months as self-reported
* Not have any history of epilepsy, stroke, moderate-to-severe traumatic brain injury or se-vere migraines
* Not have history of neurosurgery as self-reported
* Not have history of major psychiatric disorders such as schizophrenia and bipolar disorder
* Not have any other previously diagnosed disorder with symptoms similar to the TMD, such as fibromyalgia.

Exclusion Criteria:

* One absence during therapeutic sessions;

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
1. Change from baseline in Visual Analogic Scale | 14 days
  The visual analogic scale allows us to convert subjective sensations as pain on nu-merical data. A 10cm scale where 0cm is no pain and 10cm the worse imaginable pain, will be used and the subjects will be asked to mark a point on the scale repre-senting their pain. This instrument was used to compare VAS values on days 1, 5 and 10.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kijak, DSc, Study Director — Pomeranian Medical University

IPD SHARING:
Plan to Share IPD: No